CLINICAL TRIAL: NCT03449784
Title: Observatory of Patients With Dyslipidemia Hospitalized in Endocrinology-Diabetology-Nutrition Unit: Observational Study
Brief Title: Assessment of Compliance With European and French Guidelines for the Management of Dyslipidaemias
Acronym: OBDYSLIP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0104
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Patient With Dyslipidemia
Keywords: dyslipidemia; lipid-lowering therapy; cardiovascular risk; diabetes; low-density lipoprotein cholesterol
MeSH Terms: conditions — Dyslipidemias; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with dyslipidemia non achieving LDL-C target: patients with dyslipidemia non achieving LDL-C target
  Interventions: Other: Detection of patients with dyslipidemia
- patients with dyslipidemia achieving LDL-C target: patients with dyslipidemia achieving LDL-C target
  Interventions: Other: Detection of patients with dyslipidemia

INTERVENTIONS:
Other: Detection of patients with dyslipidemia — Detection of patients with dyslipidemia

SUMMARY:
Cardiovascular disease (CVD) due to atherosclerosis of the arterial vessel wall and to thrombosis is the foremost cause of premature mortality and of disability-adjusted life years in Europe, and is also increasingly common in developing countries. In the European Union, the economic cost of CVD represents annually €192 billion in direct and indirect healthcare costs. The main clinical entities are coronary artery disease (CAD), ischaemic stroke, and peripheral arterial disease (PAD). The causes of these CVDs are multifactorial. Some of these factors relate to lifestyles, such as tobacco smoking, lack of physical activity, and dietary habits, and are thus modifiable. Other risk factors are also modifiable, such as elevated blood pressure, type 2 diabetes, and dyslipidaemias, or non-modifiable, such as age and male gender. LDL-cholesterol (LDL-C) is one of the major risk factors for CVD, through its role in the development of atherosclerosis. The efficacy of statins has been demonstrated by a considerable amount of literature not only in lowering LDL cholesterol levels but also in reducing cardiovascular events, both in diabetes and non-diabetes patients. Guidelines for the management of dyslipidemia have emerged from different countries. Thereby, in 2016 the French Society of Endocrinology (SFE) and the New French Society of Atherosclerosis (NSFA) published a consensus statement on the management of dyslipidemias integrating features from European recommendations and in 2017 the Haute Autorité de Santé updated the French guidelines. However, LDL-C goal attainment has rarely been assessed specifically in diabetes population, in which CVD is of particular importance. This study aimed to assess the rate of dyslipidaemias in a population of patient hospitalized in Endocrinology-Diabetology-Nutrition unit.

This observational study was carried in the Diabetes-Nutrition unit of the University Hospital of Montpellier - France. All consecutive patients admitted to that unit during the study period were assessed for eligibility. Data on age, sex, tobacco smoking, body mass index, hypertension (treatment of previously diagnosed hypertension or blood values > 140/90 mmHg), presence and type of CVD (coronary artery disease, stroke and transient ischemic attack, peripheral arterial disease), were collected at admission. LDL-C, HDL-C and triglycerides levels calculated with the Friedewald formula, and glomerular filtration rate calculated according to the CKD-EPI formula were obtained from blood samples taken within 24 hours of hospitalization admission. Information on the name and daily dose of lipid lowering drugs (statins, fibrate, ezetimibe …) at admission was documented. Cardiovascular risk level and LDL-C target values were defined according to 2011 and 2016 ESC guidelines and 2017 French guidelines.

ELIGIBILITY:
Inclusion criteria:

- Patients aged above 18 years old, admitted to the department during the study period and hospitalized for at least 24 hours, blood samples taken within 24 hours of hospitalization admission (LDL-C, triglycerides)

Exclusion criteria:

- Patients with elevated triglycerides (>4.5 mmol/L or >400 mg/dL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population was composed of patient hospitalized in Diabetes-Nutrition unit of Montpellier University hospital.
Sampling Method: Non-Probability Sample
Enrollment: 977 (Estimated)
Dates: Start 2012-05-01 (Actual); Primary Completion 2040-11-01 (Estimated); Study Completion 2041-05-01 (Estimated)

PRIMARY OUTCOMES:
number with dyslipidemia | 1 day
  number of patient with dyslipidemia

SECONDARY OUTCOMES:
number of patient not achieving LDL-C target according to cardiovascular risk | 1 day
  number of patient not achieving LDL-C target according to cardiovascular risk

CONTACTS AND LOCATIONS:
Overall Officials: Cyril BREUKER, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Breuker C, Macioce V, Lasse A, Zogheib ML, Cavallin L, Herman F, Picot MC, Gourdy P, Sallerin B, Avignon A, Sultan A. Attainment of LDL-cholesterol target in high cardiovascular risk type 1 diabetic French people. Diabetes Metab. 2024 Nov;50(6):101568. doi: 10.1016/j.diabet.2024.101568. Epub 2024 Aug 3. PMID 39098658
- [Derived] Breuker C, Clement F, Mura T, Macioce V, Castet-Nicolas A, Audurier Y, Boegner C, Morcrette E, Jalabert A, Villiet M, Avignon A, Sultan A. Non-achievement of LDL-cholesterol targets in patients with diabetes at very-high cardiovascular risk receiving statin treatment: Incidence and risk factors. Int J Cardiol. 2018 Oct 1;268:195-199. doi: 10.1016/j.ijcard.2018.04.068. PMID 30041785